CLINICAL TRIAL: NCT00560872
Title: Randomized Controlled Study of Remote Magnetic Catheter Navigation for Cavotricuspid Isthmus Mapping and Ablation in Patients With Typical Atrial Flutter
Brief Title: Remote Magnetic Navigation For Cavotricuspid Isthmus Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Goettingen (Other)
Collaborators: Stereotaxis (Industry)
Responsible Party: PD Dr. med. Dirk Vollmann, Universitaetsmedizin Goettingen, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MN-07-022-GOE; Stereotaxis#07-022
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Atrial Flutter
Keywords: atrial flutter; ablation; navigation
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): conventional ablation with manual catheter navigation
  Interventions: Procedure: cavotricuspid isthmus ablation
- 2 (Active Comparator): ablation with remote magnetic catheter navigation
  Interventions: Device: remote magnetic catheter navigation

INTERVENTIONS:
Device: remote magnetic catheter navigation — use of the Stereotaxis system
  Arms: 2
Procedure: cavotricuspid isthmus ablation — conventional (manual) approach
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the influence of remote magnetic catheter navigation on the safety and efficacy of mapping and radiofrequency ablation of the cavotricuspid isthmus in patients with typical atrial flutter.

ELIGIBILITY:
Inclusion Criteria:

* ECG documentation of at least 1 episode of typical atrial flutter

Exclusion Criteria:

* Prior right atrial ablation
* Ferromagnetic implants that may interfere with the magnetic navigation system
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
ablation duration and fluoroscopy time | 3 months

SECONDARY OUTCOMES:
total procedure duration, success, ablation characteristics, flutter recurrence, complications | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Vollmann, PD Dr. med., Principal Investigator — Herzzentrum, Abteilung Kardiologie, Universitaetsmedizin Goettingen
Locations (1):
- Herzzentrum, Abteilung Kardiologie, Georg-August-Universitaet, Göttingen, Germany

REFERENCES:
- [Derived] Vollmann D, Luthje L, Seegers J, Hasenfuss G, Zabel M. Remote magnetic catheter navigation for cavotricuspid isthmus ablation in patients with common-type atrial flutter. Circ Arrhythm Electrophysiol. 2009 Dec;2(6):603-10. doi: 10.1161/CIRCEP.109.884411. PMID 20009074